CLINICAL TRIAL: NCT05701878
Title: Field Test of COVID-19 Self-testing With Rapid Antigen Tests
Brief Title: COVID-19 Self-testing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Yael Hirsch-Moverman, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AAAU0815
Record Dates: First submitted 2023-01-24; First posted 2023-01-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19; self-testing; mobile-app; SMARTest; randomized control trial; RCT; antigen test; mobile health; digital health
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will either be given access to the self-testing mobile app or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (App) Group (Experimental): Participants in this group will be given access to a COVID-19 self-testing app (SMARTest). Access to the app, given exclusively to this group, will be in addition to the 12 COVID-19 self-test kits participants receive.
  Interventions: Behavioral: SMARTest mobile app for COVID-19 self-testing
- Control (No App) Group (No Intervention): Participants in this group will not be given access to the COVID-19 self-testing app (SMARTest). Participants will only receive the 12 COVID-19 self-test kits.

INTERVENTIONS:
Behavioral: SMARTest mobile app for COVID-19 self-testing — The mobile app has self-testing features and information with regard to self-testing and COVID-19.
  Arms: Intervention (App) Group

SUMMARY:
The goal of this clinical trial is to understand how the introduction of an app-based intervention changes knowledge, attitudes, and practices on COVID-19 self-testing.

DETAILED DESCRIPTION:
Rapid diagnostic testing has been shown to be an important tool in controlling the spread of the COVID-19 pandemic by identifying people when they are likely to be most contagious and reducing crowding at testing sites. In addition to employer-mandated testing, rapid antigen tests are becoming increasingly used by individuals. A method to promote frequent self-testing would help break the chain of viral transmission, slow the spread of disease, slow the spread of vaccine-resistant variants, and improve pandemic management.

The ubiquity of smartphones along with their data connectivity capabilities and onboard sensors make them an attractive tool to complement rapid diagnostic tests and an important component of decentralized testing. Smartphone-based tools have shown high acceptability among healthcare workers for the real-time tracking of rapid test results.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 18 years old or older
* Owns a smartphone running either Android or iOS operating systems
* Willing to download a COVID-19 self-testing app
* Willing to receive and send text messages for the study (and fill out surveys linked from text messages)

Exclusion Criteria:

* Not willing to self-test themselves with COVID-19 rapid tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
COVID-19 Self-Testing Knowledge, Attitudes, and Practices Questionnaire Score - study initiation | Baseline
  COVID-19 Rapid Tests Knowledge, Attitudes, and Practices Questionnaire is a self-assessment measuring participant attitudes, knowledge, and practices toward COVID-19 rapid tests and self-testing.
COVID-19 Self-Testing Knowledge, Attitudes, and Practices Questionnaire Score - study completion | At study completion (About 1 month after enrollment)
  COVID-19 Rapid Tests Knowledge, Attitudes, and Practices Questionnaire is a self-assessment measuring participant attitudes, knowledge, and practices toward COVID-19 rapid tests and self-testing.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Hirsch-Moverman, PhD, Principal Investigator — Columbia University; Samuel K. Sia, PhD, Study Chair — Columbia University
Locations (1):
- ICAP Harlem Prevention Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. However if plans change and IPD is made available to other researchers, the data will be de-identified unless disclosure of the information is required by law or the participant has authorized the disclosure.
  Data that may be shared (not individual participant data) would consist of responses to the baseline and follow-up questionnaires, and recorded self-testing frequency. If the participant is in the intervention (App) group of the study, this may also include scans of the self-tests taken through the app, user engagement metrics tracked by the app, and responses to app feedback questionnaire(s). To reiterate, this data would be de-identified and would not be able to be traced back to the participant.